CLINICAL TRIAL: NCT01523899
Title: A Randomized Clinical Trial Comparing Use of Rapid Molecular Testing for Staphylococcus Aureus for Patients With Cutaneous Abscesses in the Emergency Department With Standard of Care.
Brief Title: Antimicrobial Stewardship Through MRSA Diagnosis in Emergency Department (ED) Patients With Abscesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Larissa May, Assistant Professor of Emergency Medicine, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 030927
Record Dates: First submitted 2012-01-26; First posted 2012-02-01 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Cutaneous Abscess
Keywords: SSTI; cutaneous abscess; boil
MeSH Terms: conditions — Furunculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xpert MRSA/SA SSTI (Experimental): use of the Xpert MRSA/SSTI diagnostic assay
  Interventions: Device: Xpert MRSA/SA SSTI
- Standard culture (Active Comparator): performance of standard bacterial culture of abscess material
  Interventions: Diagnostic Test: Standard culture

INTERVENTIONS:
Device: Xpert MRSA/SA SSTI — Use of Xpert MRSA/SA SSTI assay
  Arms: Xpert MRSA/SA SSTI
Diagnostic Test: Standard culture
  Arms: Standard culture

SUMMARY:
This study expands upon pilot data for feasibility since May 2011. The study aims to evaluate the effect of rapid test availability on use of targeted spectrum antibiotics for non-MRSA abscesses in ambulatory patients in the Emergency Department (ED). The multi-institutional study will assess the feasibility of providing the GeneXpert® MRSA/SA SSTI assay to the ED and evaluate the impact of delivering the test result to clinicians in real-time on patient management decisions regarding the use of antimicrobial agents. Patients are randomized to standard culture (control arm) or to the GeneXpert® assay plus standard culture.

DETAILED DESCRIPTION:
Our objective was to determine whether real-time availability of rapid molecular results of Staphylococcus aureus would impact emergency department clinician antimicrobial selection for adults with cutaneous abscesses.

We performed a prospective, randomized controlled trial in two urban emergency departments comparing a rapid molecular test with standard of care culture-based testing. Follow-up telephone calls were made at between 2 and 7 days, 1 month, and 3 months after discharge.

Patients at least 18 years old presenting with a chief complaint of abscess, cellulitis, or insect bite and receiving incision and drainage were eligible. Seven hundred seventy-eight people were assessed for eligibility and 252 met eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 years or older with community onset abscess

Exclusion Criteria:

* previous treatment for same abscess in past 14 days
* postoperative infection
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2011-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larissa S May, MD, Principal Investigator — The George Washington University
Locations (2):
- United States (2):
  - The George Washington University, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] May LS, Rothman RE, Miller LG, Brooks G, Zocchi M, Zatorski C, Dugas AF, Ware CE, Jordan JA. A Randomized Clinical Trial Comparing Use of Rapid Molecular Testing for Staphylococcus aureus for Patients With Cutaneous Abscesses in the Emergency Department With Standard of Care. Infect Control Hosp Epidemiol. 2015 Dec;36(12):1423-30. doi: 10.1017/ice.2015.202. Epub 2015 Aug 26. PMID 26306996

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Culture: Standard bacterial culture and susceptibility testing
Period: Overall Study
Arm/Group | Xpert MRSA/SA SSTI | Standard Culture
Started | 126 | 126
Completed | 126 | 126
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Culture: Xpert MRSA/SA SSTI: Use of Xpert MRSA/SA SSTI assay
- Total: Total of all reporting groups
Arm/Group | Xpert MRSA/SA SSTI | Standard Culture | Total
Number analyzed (Participants) | 126 | 126 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 126 | 252
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (13.4) | 36.5 (13.8) | 36 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 73 | 136
  Male | 63 | 53 | 116
Region of Enrollment [Number; unit: participants]
  United States | 126 | 126 | 252

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Antibiotic Usage at the Time of the ED Visit
Description: Number of Participants with Antibiotic Usage at the time of the ED visit (narrow spectrum, broad spectrum, or none) will be recorded at the time of the ED visit
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Xpert MRSA/SA SSTI | Standard Culture
Number analyzed (Participants) | 126 | 126
Participants | 97 | 96
Statistical Analysis 1: Comparison: Xpert MRSA/SA SSTI vs Standard Culture; Test type: Superiority; Pearson chi squared, Fisher exact, 2 sample t-tests; Mean Difference (Final Values) = 0.145

2. Secondary Outcome: Participant Clinical Improvement Post-treatment at One Week
Description: clinical improvement (decreasing erythema, pain, swelling, drainage, and presence or absence of fever) will be documented at 2-7 day phone follow up and 1 and 3 months
Time Frame: 2 to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Xpert MRSA/SA SSTI | Standard Culture
Number analyzed (Participants) | 103 | 103
Participants | 91 | 94
Statistical Analysis 1: Comparison: Xpert MRSA/SA SSTI vs Standard Culture; Test type: Superiority; p > 0.05, Chi-squared

3. Secondary Outcome: Clinical Outcome at One or Three Months
Description: Recurrence of abscess within a three month time period
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Xpert MRSA/SA SSTI | Standard Culture
Number analyzed (Participants) | 91 | 88
Participants | 26 | 24

ADVERSE EVENTS:
Description: Adverse events were not expected with this diagnostic study and were not monitored for this study.
Arm/Group | Xpert MRSA/SA SSTI | Standard Culture
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No